CLINICAL TRIAL: NCT07375680
Title: Evaluation of the Effect of Hemoglobin A1c Levels on Gastric Emptying Assessed by Gastric Ultrasound
Brief Title: HbA1c Levels and Gastric Emptying Assessed by Gastric Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Merve Yaman, MD,Assistant Professor of Anesthesiology, Kutahya Health Sciences University
Other Study IDs: KHSU-HbA1c-GastricUS
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Delayed Gastric Emptying; Diabetes Mellitus; Pulmonary Aspiration
Keywords: Hemoglobin A1c; Gastric Ultrasonography; General Anesthesia; Preoperative Assessment
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Adult patients scheduled for elective surgery under general anesthesia who undergo preoperative bedside gastric ultrasonography as part of an observational study.

SUMMARY:
Delayed gastric emptying increases the risk of pulmonary aspiration during general anesthesia. Diabetes mellitus and poor long-term glycemic control have been associated with impaired gastric motility. Hemoglobin A1c (HbA1c) is a marker of long-term glycemic control; however, its relationship with gastric emptying in surgical patients is not fully understood.

This prospective observational study aims to evaluate the association between HbA1c levels and gastric emptying using preoperative bedside gastric ultrasonography. Adult patients scheduled for elective surgery under general anesthesia will undergo gastric ultrasound examination after standard fasting. Gastric antral cross-sectional area and estimated gastric volume will be assessed and compared according to HbA1c levels.

The findings of this study may help improve preoperative risk stratification for aspiration and support individualized anesthetic management in patients with impaired glycemic control.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate the relationship between hemoglobin A1c (HbA1c) levels and gastric emptying in adult surgical patients using bedside gastric ultrasonography.

Adult patients aged 18 to 70 years, scheduled for elective surgery under general anesthesia, will be enrolled. After standard preoperative fasting according to current guidelines, all participants will undergo a preoperative gastric ultrasound examination performed by a trained anesthesiologist. The gastric antrum will be assessed in standardized positions, and the antral cross-sectional area will be measured. Estimated gastric volume will be calculated using validated ultrasound-based formulas.

HbA1c levels will be obtained from preoperative laboratory records, and patients will be analyzed according to their HbA1c values. Gastric ultrasound findings, including antral cross-sectional area and estimated gastric volume, will be compared across different HbA1c levels.

Demographic data, anthropometric measurements including body mass index and waist circumference, fasting duration, and relevant clinical characteristics will also be recorded. The primary objective is to assess the association between HbA1c levels and gastric emptying parameters. Secondary analyses will explore potential factors associated with delayed gastric emptying.

The results of this study may contribute to improved preoperative risk assessment for pulmonary aspiration and support individualized anesthetic management in patients with impaired glycemic control.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 70 years. ASA physical status I-III. Scheduled for elective surgery under general anesthesia. Ability to provide written informed consent.

Exclusion Criteria:

Scheduled for emergency surgery. Refusal or inability to provide informed consent. Pregnancy. Age <18 years or >70 years. History of gastric surgery. Neuromuscular disease. Current use of opioid or anticholinergic medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 70 years scheduled for elective surgery under general anesthesia at a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying assessed by gastric ultrasound | The preoperative period,immediately before induction of anesthesia
  Gastric emptying will be assessed preoperatively using bedside gastric ultrasonography by measuring gastric antrum cross-sectional area and estimating gastric volume with validated ultrasound-based methods.

CONTACTS AND LOCATIONS:
Overall Officials: merve yaman, MD, Assistant Professor, Principal Investigator — Kutahya Health Science University; emine gök, MD, Study Director — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University Training and Research Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No